CLINICAL TRIAL: NCT02977520
Title: Preoperative Assessment and Individualized Operation Optimization of Acute Ruptured Cerebral Aneurysms
Acronym: PAOCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TWKY-2016-ZD-01-10
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Printing, Three-Dimensional, Simulation Training
MeSH Terms: interventions — Printing, Three-Dimensional

ARMS (2):
- Interventional group (Experimental): Obtain the CTA data of cerebral aneurysms and built the 3D printing models. Combined with the 3D model, the neurosurgeon can complete the discussion of preoperative prediction of aneurysms and recognize the adjacent bone, blood vessels, aneurysm directions and so on. In addition, the model can also be used to the young doctor's training, and the patient and their families can be convenient and intuitive understanding of the disease, so as to form a good communication between doctors and patients.
  Interventions: Procedure: Printing, Three-Dimensional
- general group (No Intervention): Obtain the CTA data of cerebral aneurysms, the neurosurgeon complete the discussion of preoperative prediction of aneurysms.

INTERVENTIONS:
Procedure: Printing, Three-Dimensional — To establish 3D model of cerebral aneurysms and have preoperative evaluation.
  Arms: Interventional group

SUMMARY:
Cerebral aneurysm is one of the main diseases that seriously affect human health. The most important treatment method is surgical clipping and endovascular embolization. Not complete occlusion of the aneurysm is a main risk of recurrence and rebleeding after treatment. This study is focused on the 3D model of cerebral aneurysms and preoperative evaluation. Combined with the 3D model, the neurosurgeon can complete the discussion of preoperative prediction of aneurysms and recognize the adjacent bone, blood vessels, aneurysm directions and so on. In addition, the model can also be used to the young doctor's training, and the patient and their families can be convenient and intuitive understanding of the disease, so as to form a good communication between doctors and patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years-80 years;
* Hunt-Hess grade: 0-4;
* Without other stroke, brain trauma and other neurological disease;
* Without cerebral hernia;
* Cystic aneurysm.

Exclusion Criteria:

* Age: less than 18 years or above 80 years;
* Hunt-Hess grade is 5;
* With serious previous disorder of multiple organ;
* Acute cerebral hernia;
* Aneurysms were fusiform or serpentine expansion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
time of operation | 1 to 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Luhe hospital, Beijing, Beijing Municipality, China